CLINICAL TRIAL: NCT04816344
Title: The Frequency of Emergence Delirium in Children Undergoing Outpatient Anaesthesia for Magnetic Resonance Imaging
Brief Title: Emergence Delirium in Children for Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Derya Karasu, MD, Assoc Prof., Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: U1111-1265-0994
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Delirium; Pediatric Disorder; Anesthesia
Keywords: MRI scans; pediatric; delirium; anaesthesia
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group MP (n=35): The patients were separated into four groups according to the anaesthetic agents given.
  Premedication was applied as intranasal 0.2 mg/kg midazolam, then 1 mg/kg of propofol iv bolus as an anaesthetic agent was administered, and if necessary propofol 0.5 mg/kg iv was given as additional dosage.
  Interventions: Procedure: Outpatient Anesthesia
- Group MK (n=35): Premedication was applied as intranasal 0.2 mg/kg midazolam, then 1 mg/kg ketofol (10% ketamine + 10% propofol) iv bolus as an anaesthetic agent was administered, and if necessary 0.5 mg/kg iv ketofol was given as additional dosage.
  Interventions: Procedure: Outpatient Anesthesia
- Group DP (n=35): Premedication was applied as intranasal 1 mcg/kg dexmedetomidine, then 1 mg/kg of propofol iv bolus as an anaesthetic agent was administered, and if necessary propofol 0.5 mg/kg iv was given as additional dosage.
  Interventions: Procedure: Outpatient Anesthesia
- Group DK (n=35): Premedication was applied as intranasal 1 mcg/kg dexmedetomidine, then 1 mg/kg ketofol iv bolus as an anaesthetic agent was administered, and if necessary 0.5 mg/kg ketofol iv was given as an additional dosage.
  Interventions: Procedure: Outpatient Anesthesia

INTERVENTIONS:
Procedure: Outpatient Anesthesia — The inclusion criteria were children aged between 2 and 10 years, undergoing outpatient anaesthesia for elective MRI under sedation, and classified as American Society of Anesthesiologists (ASA) grade I-II. The study exclusion criteria were defined as difficult airway, allergies to the study drugs, asthma, severe central nervous system disease (eg, brain tumour, uncontrolled seizures), mental motor retardation, the application of another procedure after MRI sedation, and those whose parents declined to participate in the study.

SUMMARY:
Sedation or anaesthesia is necessary to be able to perform magnetic resonance imaging (MRI) on children who cannot keep still or are uncooperative, and thus the targets of maximum patient safety, successful imaging, and the highest imaging quality can be achieved. There are various drugs for sedation in MRI. A child with Anaesthesia Emergence Delirium (AED) has a state of consciousness which can be described as "irritable, uncompromising, inconsistent, crying inconsistently, wailing, and kicking". The incidence of AED worldwide has been reported to vary between 18% and 80%, depending on the diagnostic criteria used. This difference can usually be explained by the use of different scales and defining criteria. In 2004, Sikich and Lerman developed the Paediatric Anaesthesia Emergence Delirium (PAED) scale, including cognitive evaluation components in addition to agitation behaviours, and the validity and reliability of this scale have been proven. In a study of anaesthesia early delirium in children by Bong et al.7 a score of ≥10 on the PAED scale was shown to have the greatest sensitivity and specificity for the diagnosis of anaesthesia early delirium.

The aim of this study was to investigate the effect on the occurrence of emergence delirium, and recovery, of propofol and ketofol in paediatric patients undergoing diagnostic MRI following premedication with intranasal dexmedetomidine and midazolam.

DETAILED DESCRIPTION:
This was a prospective, observational, and single-center study conducted between July-November 2018. The study protocol was approved by the Local Ethics Committee. The study was conducted in accordance with the principles of the Declaration of Helsinki. Written informed consent was obtained from the parent.

The patients were separated into four groups according to the anaesthetic agents given.Intranasal premedication was applied to all the patients, then an intravenous cannula was placed and the anaesthetic agents were administered intravenously. The Ramsay Sedation Scale (RSS) was used to evaluate the level of sedation, with a target of 5 points. The RSS is scored from 1-6 as follows: 1: the patient is worried and anxious, or restless, 2: the patient is calm and co-operative, and can be directed, 3: the patient only responds to instructions, 4: the patient responds rapidly to painful stimuli, 5: the patient demonstrates a slow response to painful stimuli, 6: the patient does not respond. When RSS 5 was reached following the first bolus dose of the drug, an additional dose was administered. When RSS 5 was obtained and hemodynamic stability was ensured, the patient was placed on the MRI table.

The patient was monitored in the recovery room for regaining consciousness for up to 30 mins after the procedure. AED was evaluated using the PAED scale by a nurse trained in the use of this scale. PAED scoring was repeated every 5 mins until the patient was discharged from the recovery room. If the PAED score was ≥10, a diagnosis of AED was made. Adverse events such as laryngospasm, desaturation (SpO2 <95%), respiratory depression, bradycardia, allergy, hiccoughs, nystagmus, nausea, and vomiting were recorded. When a Modified Aldrete Score of >9 was obtained, the child was observed for a further 15 mins then transferred from the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 2 and 10 years,
* undergoing outpatient anaesthesia for elective MRI under sedation,
* classified as American Society of Anesthesiologists (ASA) grade I-II.

Exclusion Criteria:

* difficult airway,
* allergies to the study drugs,
* asthma,
* severe central nervous system disease (eg, brain tumour, uncontrolled seizures),
* mental motor retardation,
* the application of another procedure after MRI sedation,
* whose parents declined to participate in the study.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children undergoing outpatient anaesthesia for elective MRI under sedation
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
emergence delirium | until 30 minutes after arrival in the recovery room
  the incidence of emergence delirium

SECONDARY OUTCOMES:
adverse events | up to 1 hour after anesthesia
  apnea, falling in saturation, increased secretin, atropine requirement, bradycardia, nausea-vomiting,hiccup

CONTACTS AND LOCATIONS:
Overall Officials: Derya Karasu, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences Turkey, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided